CLINICAL TRIAL: NCT00105820
Title: Well-being Among Veterans Enhancement Study (WAVES)
Brief Title: Evaluation Study of TIDES Depression Care Quality Improvement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MHI 99-375
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Major Depression; PTSD
Keywords: Evaluation; Quality improvement; Cluster randomized trial; Care model; Collaborative care; Informatics
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: System level depression care quality improvement

INTERVENTIONS:
Procedure: System level depression care quality improvement

SUMMARY:
In spite of the impact on veteran�s health status and treatment cost, depression is under-diagnosed and under-treated. The goal of this study is to learn how to implement a previously tested, effective collaborative care model for improving the quality of depression care across multiple Veterans Integrated Service Networks (VISNs). To achieve this goal, we are conducting a randomized controlled trial of evidence-based quality improvement (EBQI), a dissemination method that relies on expert design and local implementation of evidence-based practice interventions. We hypothesize that EBQI will result in increased rates of assessment and appropriate management of depression. Results will be useful in designing realistic chronic care programs and performance measures for continuing care improvement.

DETAILED DESCRIPTION:
Objectives: Our primary objective is to evaluate whether collaborative care EBQI results in increased rates of assessment and appropriate management of depression and decreased depressive symptomatology for veterans. Our secondary objective is to evaluate the effect of EBQI on organizational outcomes.

Methods: Three VISNs, 10, 16 and 23, are participating. Three primary care clinics within each VISN are randomized, two to the intervention and one to usual care, for a total of nine study sites. In the intervention clinics, VA leadership, assisted by study staff, tailor and implement a depression care program for patient assessment, patient self-management support, provider education, primary and mental health collaboration, and care management. The usual care clinics participate only in the evaluation. Patient recruitment is through a telephone interview. Patients who are at risk for major depression are recruited, 67 from each site. Patient outcomes including depression symptom severity on the PHQ-9 and the VA SF-12 are being assessed by telephone at six months post enrollment. Other outcome variables are adequacy of antidepressant trials, psychotherapy and specialty care visits, and treatment adherence. A utilization and cost analysis will be conducted. VISN and VAMC leadership are surveyed to assess organizational outcomes. Data is being collected through VA administrative databases, patient and staff interviews, and study records. Power calculations and data analysis planning reflect the clustered sample design.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a pt in the VA Healthcare System
* screens positive for major depression
* has a scheduled visit at a primary care site taking part in the study

Exclusion Criteria:

* severe alcohol abuse
* psychosis
* dementia
* acutely suicidal (at screening)
* lack of access to or ability to use a phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2003-06; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
At set time points the following will be measured: Recovery from depression Patient quality of life 1 year before and after: Clinic depression treatment utilization and costs

SECONDARY OUTCOMES:
Adherence to appropriate treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edmund F. Chaney, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Lisa V. Rubenstein, MD MSPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (3):
- United States (3):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Felker BL, Barnes RF, Greenberg DM, Chaney EF, Shores MM, Gillespie-Gateley L, Buike MK, Morton CE. Preliminary outcomes from an integrated mental health primary care team. Psychiatr Serv. 2004 Apr;55(4):442-4. doi: 10.1176/appi.ps.55.4.442. PMID 15067160
- [Result] Kanter JW, Epler AJ, Chaney EF, Liu CF, Heagerty P, Lin P, Felker B, Hedrick SC. Comparison of 3 Depression Screening Methods and Provider Referral in a Veterans Affairs Primary Care Clinic. Prim Care Companion J Clin Psychiatry. 2003 Dec;5(6):245-250. doi: 10.4088/pcc.v05n0601. PMID 15213794
- [Result] Felker BL, Chaney E, Rubenstein LV, Bonner LM, Yano EM, Parker LE, Worley LL, Sherman SE, Ober S. Developing effective collaboration between primary care and mental health providers. Prim Care Companion J Clin Psychiatry. 2006;8(1):12-6. doi: 10.4088/pcc.v08n0102. PMID 16862248
- [Result] Fortney JC, Steffick DE, Burgess JF Jr, Maciejewski ML, Petersen LA. Are primary care services a substitute or complement for specialty and inpatient services? Health Serv Res. 2005 Oct;40(5 Pt 1):1422-42. doi: 10.1111/j.1475-6773.2005.00424.x. PMID 16174141
- [Result] Chaney E, Rabuck LG, Uman J, Mittman DC, Simons C, Simon BF, Ritchie M, Cody M, Rubenstein LV. Human subjects protection issues in QUERI implementation research: QUERI Series. Implement Sci. 2008 Feb 15;3:10. doi: 10.1186/1748-5908-3-10. PMID 18279507
- [Result] Campbell DG, Felker BL, Liu CF, Yano EM, Kirchner JE, Chan D, Rubenstein LV, Chaney EF. Prevalence of depression-PTSD comorbidity: implications for clinical practice guidelines and primary care-based interventions. J Gen Intern Med. 2007 Jun;22(6):711-8. doi: 10.1007/s11606-006-0101-4. PMID 17503104
- [Result] Liu CF, Bolkan C, Chan D, Yano EM, Rubenstein LV, Chaney EF. Dual use of VA and non-VA services among primary care patients with depression. J Gen Intern Med. 2009 Mar;24(3):305-11. doi: 10.1007/s11606-008-0867-7. Epub 2008 Dec 20. PMID 19101777
- [Result] Waltz TJ, Campbell DG, Kirchner JE, Lombardero A, Bolkan C, Zivin K, Lanto AB, Chaney EF, Rubenstein LV. Veterans with depression in primary care: provider preferences, matching, and care satisfaction. Fam Syst Health. 2014 Dec;32(4):367-77. doi: 10.1037/fsh0000071. Epub 2014 Aug 4. PMID 25090611
- [Result] Lombardero A, Campbell DG, Harris KJ, Chaney EF, Lanto AB, Rubenstein LV. Prevalence and correlates of smoking status among veterans affairs primary care patients with probable major depressive disorder. Addict Behav. 2014 Mar;39(3):538-45. doi: 10.1016/j.addbeh.2013.10.030. Epub 2013 Nov 4. PMID 24290879
- [Result] Bolkan CR, Bonner LM, Campbell DG, Lanto A, Zivin K, Chaney E, Rubenstein LV. Family involvement, medication adherence, and depression outcomes among patients in veterans affairs primary care. Psychiatr Serv. 2013 May 1;64(5):472-8. doi: 10.1176/appi.ps.201200160. PMID 23370463
- [Result] Bonner LM, Lanto AB, Bolkan C, Watson GS, Campbell DG, Chaney EF, Zivin K, Rubenstein LV. Help-seeking from clergy and spiritual counselors among veterans with depression and PTSD in primary care. J Relig Health. 2013 Sep;52(3):707-18. doi: 10.1007/s10943-012-9671-0. PMID 23297184
- [Result] Yano EM, Chaney EF, Campbell DG, Klap R, Simon BF, Bonner LM, Lanto AB, Rubenstein LV. Yield of practice-based depression screening in VA primary care settings. J Gen Intern Med. 2012 Mar;27(3):331-8. doi: 10.1007/s11606-011-1904-5. PMID 21975821
- [Result] Zivin K, Campbell DG, Lanto AB, Chaney EF, Bolkan C, Bonner LM, Miller EM, Valenstein M, Waltz TJ, Rubenstein LV. Relationships between mood and employment over time among depressed VA primary care patients. Gen Hosp Psychiatry. 2012 Sep-Oct;34(5):468-77. doi: 10.1016/j.genhosppsych.2012.05.008. Epub 2012 Jul 6. PMID 22771108
- [Result] Chaney EF, Rubenstein LV, Liu CF, Yano EM, Bolkan C, Lee M, Simon B, Lanto A, Felker B, Uman J. Implementing collaborative care for depression treatment in primary care: a cluster randomized evaluation of a quality improvement practice redesign. Implement Sci. 2011 Oct 27;6:121. doi: 10.1186/1748-5908-6-121. PMID 22032247